CLINICAL TRIAL: NCT02310620
Title: Computer Games to Prevent Mild Cognitive Impairment and Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Gábor Csukly, Assistant Professor, Semmelweis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: M3W2012
Record Dates: First submitted 2014-12-02; First posted 2014-12-08 (Estimated); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cognitive Training (Experimental)
  Interventions: Behavioral: Cognitive training

INTERVENTIONS:
Behavioral: Cognitive training — regular playing with the logic games developed in the framework of the M3W (Mental Wellness Toolset) project (https://m3w-project.eu/)

SUMMARY:
The aim of the study is to show that regular playing with the logic games developed in the framework of the M3W (Mental Wellness Toolset) project (https://m3w-project.eu/) can prevent mild cognitive impairment (MCI) and dementia.

The secondary aim of the study is to find correlations between the results of the games and the standard assessments for dementia and MCI screening such as the Rey Verbal Learning Test.

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* Older than 50 years of age

Exclusion Criteria:

* Subjects with history of head trauma, epilepsy or stroke.
* Diagnosis of schizophrenia
* Acute manic episode

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2012-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Conversion to Mild Cognitive Impairment (?CI) (Proportion of participants who develop MCI after 3 years) | 3 years
  Proportion of participants who develop MCI after 3 years
Conversion to dementia (Proportion of participants who develop dementia after 3 years) | 3 years
  Proportion of participants who develop dementia after 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry and Psychotherapy, Budapest, Hungary